CLINICAL TRIAL: NCT02785107
Title: Facilitating an Exercise Habit Via the Multi-Process Action Control Model: A Randomized-Controlled Trial
Brief Title: Exercise Habit and M-PAC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Victoria (Other)
Responsible Party: Principal Investigator, Navin Kaushal, PhD, University of Victoria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-306
Record Dates: First submitted 2016-05-11; First posted 2016-05-27 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Public Health
Keywords: Exercise; Habit; MVPA; M-PAC; Automaticity; Physical Activity
MeSH Terms: conditions — Motor Activity; Habits

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Those who were randomized into the intervention group attended a workshop where the PI delivered a presentation that focused on establishing a preparatory exercise habit by using the M-PAC approach and proposed habit model. Participants were then provided with instructions on completing their exercise plan sheet.
  Interventions: Behavioral: M-PAC Group
- Control (No Intervention): Participants exercised on their own without receiving any instructions.

INTERVENTIONS:
Behavioral: M-PAC Group — Participants attended a workshop, completed a worksheet and received a booster phone call follow-up at week four.
  Arms: Intervention

SUMMARY:
The promotion of physical activity (PA) is paramount to public health, yet interventions in the social cognitive tradition have yielded negligible improvements. Two reasons for these results may be the over reliance on intention as the proximal determinant of behaviour and a lack of consideration of implicit/automatic determinants of PA. The purpose of this study was to apply Multi-Process Action Control (M-PAC), a framework centered on PA intention-translation and the gradual building of habit to examine PA change using a two-arm parallel design, randomized controlled trial.

DETAILED DESCRIPTION:
Background: Two of the most prominent limitations of traditional social cognitive models used to understand moderate-to-vigorous physical activity (MVPA) are the gap between intention and behaviour and the lack of consideration of implicit processes in behavioural enactment. Thus, new models are now being examined that attempt to consider these potential limitations. Multi-Process Action Control (M-PAC) is one such attempt to build a more comprehensive schematic, whereby intention is established via the means of constructs from traditional social cognitive theories (i.e., outcome expectations, perceived capability), but the success of translating this intention to behaviour depends on behavioural-regulation (self-regulatory tactics) (BR), affective judgments (expected pleasure) (AJ) and opportunity (time, access). Over time, M-PAC proposes that habit (stimulus -behaviour bonds) and identity (role-behaviour bonds) develop from performing the behaviour and largely contribute to the maintenance of PA.

Aim: The purpose of this study was to conduct at two-arm parallel design, RCT to determine if the M-PAC experimental group would demonstrate greater change in PA and post-intention constructs across time.

Methods: Participants (n=94) were inactive new gym members and were randomized into a control or M-PAC experimental group. The experimental group attended a workshop and received a booster phone call follow-up at week four. Measures for both groups included accelerometry and M-PAC at baseline and at week eight.

ELIGIBILITY:
Inclusion Criteria:

* New gym member
* age 18-65
* Par-Q pass

Exclusion Criteria:

* age <18 or 65+
* Par-Q fail

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
GT3X+ Actigraph Activity Monitors (for measuring physical activity) | Baseline to week eight
  Participants wear accelerometers for one week at baseline and at week eight to record their physical activity.

SECONDARY OUTCOMES:
Self-Report Behavioural Automaticity Index (self report, survey question) | Baseline, week four, week eight
  The Self-Report Behavioral Automaticity Index (SRBAI) was used to assess preparatory habit. The SRBAI consists of 4 items on a 5-point Likert scale with 1 being strongly disagree to 5 being strongly agree. The question stem stated ''When I prepare to exercise…'' which was then followed by four items on the scale: ''I do it without having to consciously remember'', ''I do it automatically'', ''I do it without thinking'', and ''I start before I realize I am doing it''.

OTHER OUTCOMES:
Environmental Cues (self report, survey question) | Baseline, week four, week eight
  The following item was used to assess if participants implemented the use of cues: "I use cues at home to remind me to exercise (e.g. placing a water bottle on my desk or gym clothes on the bed). The item was rated on a five point Likert scale which ranged from "1=strongly disagree" to "5= strongly agree".
Temporal Consistency (self report, survey question) | Baseline, week four, week eight
  The item was worded "How consistently do you exercise at the same time each day? (e.g., exercising every morning at 7 am, or exercising daily after supper)". The question was asked on a five point Likert scale which range from "1=not consistent at all" to "5=very consistent".

CONTACTS AND LOCATIONS:
Overall Officials: Navin Kaushal, PhD, Principal Investigator — University of Victoria
Locations (1):
- University of Victoria, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaushal N, Rhodes RE, Spence JC, Meldrum JT. Increasing Physical Activity Through Principles of Habit Formation in New Gym Members: a Randomized Controlled Trial. Ann Behav Med. 2017 Aug;51(4):578-586. doi: 10.1007/s12160-017-9881-5. PMID 28188586